CLINICAL TRIAL: NCT01842685
Title: Bladder Thermal Distention for Patients With Refractory Overactive Bladder
Acronym: OAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 216/12
Record Dates: First submitted 2013-04-14; First posted 2013-04-30 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Bladder Distention
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bladder Thermal Distention (Experimental): Continuous irrigation of the bladder with warm saline (up to 45 Celsius) using a specific 3 ways catheter. The procedure will last 1 hour. Saline will be irrigated by the PelvixTT system.
  Interventions: Procedure: Bladder Thermal Distention

INTERVENTIONS:
Procedure: Bladder Thermal Distention — Bladder Thermal Distention is an approved procedure in Europe from 2006. The treatment is hydrodistention of the bladder with a warm saline (up to 45C). The procedure lasts 1 hour. The saline is infused constantly through a 3 ways specific catheter (Unithermia 18F) by the PelvixTT system.
  Other Names: PelvixTT - Hyperthermia Elmedical LTD, Israel

SUMMARY:
In this study, the investigators will evaluate the efficacy of Bladder Thermal Distention (BTD) in patients with overactive bladder syndrome who failed previous treatment of anticholinergic drugs.

The investigators' hypothesis is that it will improve the storage symptoms.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Patients with overactive bladder syndrome
2. Detrusor Overactivity proven in urodynamic test

Exclusion criteria:

1. Mixed urinary incontinence
2. Active urinary tract infection
3. Urethral Stricture

Outcome measures:

1. Bladder Diaries
2. Urgency questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Patients with overactive bladder syndrome
* Detrusor Overactivity proven in urodynamic test

Exclusion criteria:

* Mixed urinary incontinence
* Active urinary tract infection
* Urethral Stricture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Urgency Questionnaire | up to 1 year
  Patients will complete the validated USIQ questionnaire

SECONDARY OUTCOMES:
Daily frequency of micturitions on Bladder Diary | up to 1 year
  Patients will complete bladder diaries before and after the procedure. Frequencies of micturitions per day will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Kobi Stav, MD, Principal Investigator — Assaf Harofe MC
Locations (1):
- Assaf Harofe MC, Tel Aviv Region, Zeriffin, Israel